CLINICAL TRIAL: NCT00148278
Title: Prospective, Multicenter, Randomized, Double-Blind Study Comparing Safety and Efficacy of Norepinephrine Plus Dobutamine Versus Epinephrine Alone in Septic Shock.
Brief Title: Norepinephrine Plus Dobutamine Versus Epinephrine Alone for the Management of Septic Shock
Acronym: CATS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Djillali Annane, Assistance Publique Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFSSAPS 990931; AOM97123; CIC0203/001
Record Dates: First submitted 2005-09-01; First posted 2005-09-07 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Septic Shock; Severe Sepsis; Infections
Keywords: Catecholamines; Septic shock
MeSH Terms: conditions — Shock, Septic; Sepsis; Infections | interventions — Norepinephrine; Dobutamine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): norepinephrine plus dobutamine
  Interventions: Drug: norepinephrine and dobutamine
- 2 (Active Comparator): epinephrine
  Interventions: Drug: epinephrine plus placebo of dobutamine

INTERVENTIONS:
Drug: norepinephrine and dobutamine — continuous infusion of norepinephrine titrated to maintain a mean arterial pressure at 70mmHg or more and dobutamine could be added as a continuous infusion when cardiac index was of less than 2.5 liters per squared meter of body surface
  Arms: 1
Drug: epinephrine plus placebo of dobutamine — epinephrine was titrated to maintain a mean arterial pressure at 70mmHg or more and placebo of dobutamine was titrated in case of a cardiac index lower than 2.5 liters per squared meters of body surface
  Arms: 2

SUMMARY:
Catecholamines infusion is a major component of septic shock management. International guidelines recommend that norepinephrine should be preferred to epinephrine, though phase III trials are lacking. The present study aimed at comparing the efficacy and safety of norepinephrine plus dobutamine to that of epinephrine in adults with septic shock.

DETAILED DESCRIPTION:
The french Conference on Consensus on catecholamines use in septic shock has underlined the importance of carrying out a clinical trial to clarify the use of epinephrine, norepinephrine and dobutamine in the management of multiple organ failure associated with severe sepsis. The main objective of the study was therefore to compare the effects of the combination of dobutamine and norepinephrine to those of epinephrine alone in patients with septic shock. In this purpose, patients were randomly assigned to receive either epinephrine or norepinephrine plus dobutamine and drugs were titrated to maintain blood pressure over 70 mmHg. Main outcome was 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* Informed consent

Presenting from less than 7 days :

* One or more infectious site
* At least 2 of the following criteria: temperature > 38°C or < 36.5°C, respiratory rate > 20 breaths per min or PaCO2 < 32 mmHg or mechanical ventilation, heart rate > 90 beats/min, white blood cell count > 12,000/mm3 or < 4,000/mm3
* At least 2 of the following criteria: PaO2/FiO2 ratio <280 mmHg (if mechanical ventilation, urinary output of less than 0.5 mL/kg of body weight or < 30 mL/h at least 1 hour, plasma lactate > 2 mmol/L, platelet count < 100,000 /mm3

And presenting from at least 24 hours:

* Systolic blood pressure < 90 mmHg or mean blood pressure < 70 mmHg (for at least 30 min);
* 1000 mL fluid replacement or pulmonary capillary wedge pressure > 12 mmHg
* Dopamine infusion at 15 µg/kg/min for at least 1 hour, or epinephrine or norepinephrine in first intention

Exclusion Criteria:

* Pregnant woman
* Obstructive cardiomyopathy
* Acute coronary disease
* Non infectious shock
* Care limitation
* White blood cell count < 500 /mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 1999-10; Primary Completion 2004-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
28 Day mortality | 28 Day

SECONDARY OUTCOMES:
-28-day survival distribution | Day 28
-Survival rate at days 14, 28, 90, 6 months and 1 year. | one year
-Rate of patients with secondary care limitation | one year
-Organ failure between randomization and day 28. | Day 28
-Serious adverse events between randomization and exit of intensive care unit. | one year
-Onset of a reversible clinical event between randomization and exit of intensive care unit (bronchospasm, cutaneous rash, tachycardia) | one year
-Time on vasopressors | Day 90
-Time in intensive care unit | one year
-Time in hospital | one year
-Costs | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD, PhD, Study Director — Assistance Publique Hôpitaux de Paris - University of Versailles; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (15):
- France (15):
  - Réanimation Médicale - Hôpital Louis Mourier, Colombes
  - Réanimation Polyvalente - Hôpital de Corbeil, Corbeil
  - Service de Réanimation Médicale - Hôpital Poincaré, Garches
  - Réanimation Médicale - Hôpital André Mignot, Le Chesnay
  - Réanimation Polyvalente - Hôpital Dupuytren, Limoges
  - Réanimation Polyvalente - Hôpital Nord, Marseille
  - Réanimation Chirurgicale - Hôpital Central, Nancy
  - Service de Réanimation Médicale - Hôpital Central, Nancy
  - Service d'anesthésiologie - HIA Val de Grâce, Paris
  - Réanimation Médicale - Hôpital Saint Louis, Paris
  - Réanimation Polyvalente - Hôpital Saint Joseph, Paris
  - Réanimation Médicale - Hôpital Georges Pompidou, Paris
  - Réanimation Médicale - CHI de Poissy, Poissy
  - Réanimation - CH Victor Provo, Roubaix
  - Réanimation Polyvalente - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Annane D, Vignon P, Renault A, Bollaert PE, Charpentier C, Martin C, Troche G, Ricard JD, Nitenberg G, Papazian L, Azoulay E, Bellissant E; CATS Study Group. Norepinephrine plus dobutamine versus epinephrine alone for management of septic shock: a randomised trial. Lancet. 2007 Aug 25;370(9588):676-84. doi: 10.1016/S0140-6736(07)61344-0. PMID 17720019